CLINICAL TRIAL: NCT04185584
Title: A Long-Term Safety Follow-Up Study of SCM AGH in Subjects Who Participated in the ADT2002 Study
Brief Title: Long-Term Safety Follow-Up Study of SCM-AGH in Subjects Who Participated and Administered SCM-AGH in to Severe Atopic Dermatitis Clinical Trials
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SCM Lifescience Co., LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADT2002-LTFU
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dermatitis, Atopic
Keywords: SCM-AGH; Atopic Dermatitis; Stem cell therapy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not Applicable (Observational Study) — Not Applicable (Observational Study)

SUMMARY:
This is a long-term safety follow-up study of the Phase I/II multicenter study of SCM-AGH in subjects with moderate to severe atopic dermatitis. subjects will be followed up for a maximum period of 240 weeks after the first dose of investigational product. Only subjects previously enrolled in protocol ADT2002 (ClinicalTrials.gov ID: NCT04179760) will be eligible for this long-term follow-up protocol.

DETAILED DESCRIPTION:
Subjects who meet all eligibility criteria for Long Term Follow Up(LTFU) study participation at the ADT2002 End of Treatment(EOT) visit may continue LTFU for a maximum period of up to 240 weeks post first dose of investigational product. No additional dosing will be administered on this LTFU protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide written informed consent
2. Subjects who have received at least 1 dose of SCM-AGH in the ADT2002 study
3. Subjects who are willing to comply with the visit schedule and study requirements for reporting relevant information to the site.

Exclusion Criteria:

1. Subjects who are unable to comply with the visit schedule prior to Week 240 after first dose of SCM AGH

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received at least 1 dose of SCM-AGH in the ADT2002 study (ClinicalTrials.gov ID: NCT04179760)
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety assessment of SCM-AGH in subjects with moderate to severe Atopic Dermatitis(AD) | Up to 5 Years
  Number of occurrence of treatment-related adverse events (≥ Grade 3 in severity (NCI-CTCAE, v5.0))
Long-term concomitant medication assessment of SCM-AGH in subjects with moderate to severe Atopic Dermatitis(AD) | Up to 5 Years
  Number of occurrence of use of medications related to adverse events

SECONDARY OUTCOMES:
Outcome of unresolved Adverse Events(AEs) from ADT2002 study | Up to 5 Years
Clinically important physical examination findings | Up to 5 Years
  Number of abnormality in general appearance, skin, eyes/ears/nose/throat, head and neck, cardiovascular, respiratory, abdomen, extremities, lymph nodes, musculoskeletal and neurologic.
Number of occurrence of Abnormal, clinically significant in hematology laboratory results | Up to 5 Years
  Hematology panel: alkaline phosphatase [ALP], blood urea nitrogen, creatinine, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), albumin, total protein, total bilirubin, uric acid, glucose, cholesterol, sodium, potassium, chloride, calcium, phosphorus
Number of occurrence of Abnormal, clinically significant in chemistry laboratory results | Up to 5 Years
  Chemistry panel: hemoglobin, hematocrit, red blood cells, white blood cells (WBC), WBC differential count, platelets
Number of occurrence of Abnormal, clinically significant in urinalysis laboratory results | Up to 5 Years
  Urinalysis panel: specific gravity (SG), color, pH, protein, glucose, bilirubin, blood, WBC

CONTACTS AND LOCATIONS:
Overall Officials: Gwang Seong Choi, MD-Ph.D, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea